CLINICAL TRIAL: NCT02754856
Title: Pilot Study Assessing the Safety and Tolerability of the Neoadjuvant Use of Tremelimumab (Anti-CTLA-4) Plus Durvalumab (MEDI4736) (Anti-PD-L1) in the Treatment of Resectable Colorectal Cancer Liver Metastases
Brief Title: Tremelimumab and Durvalumab in Treating Patients With Colorectal Cancer With Liver Metastases That Can Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0828; NCI-2016-00772 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0828 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-04-26; First posted 2016-04-28 (Estimated); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Carcinoma in the Liver; Resectable Mass; Stage IV Colorectal Cancer AJCC v7; Stage IVA Colorectal Cancer AJCC v7; Stage IVB Colorectal Cancer AJCC v7
MeSH Terms: conditions — Colorectal Neoplasms | interventions — durvalumab; Immunoglobulin G; Disulfides; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tremelimumab, durvalumab) (Experimental): Patients receive tremelimumab IV over 1 hour and durvalumab IV over 4 hours during week 11. Between weeks 15 and 17, patients undergo liver surgery. Patients then receive durvalumab IV over 1 hour during weeks 21, 25, 29, and 33.
  Interventions: Biological: Durvalumab; Other: Laboratory Biomarker Analysis; Procedure: Therapeutic Conventional Surgery; Biological: Tremelimumab

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Therapeutic Conventional Surgery — Undergo liver surgery
Biological: Tremelimumab — Given IV
  Other Names: Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP-675; CP-675,206; CP-675206; Ticilimumab

SUMMARY:
This phase I trial studies the side effects and how well tremelimumab and durvalumab work in treating patients with colorectal cancer that has spread to the liver and can be removed by surgery. Immunotherapy with monoclonal antibodies, such as tremelimumab and durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety and feasibility of adding tremelimumab 75 mg intravenously (IV) plus durvalumab (MEDI4736) 1500 mg administered once pre-operatively and 4 cycles of durvalumab 1500 mg IV every 4 weeks for 4 cycles post-operatively in patients who are candidates for resection for colorectal cancer liver metastases.

SECONDARY OBJECTIVES:

I. Explore the changes in various immune parameters, including programmed cell death-1 ligand 1 (PD-L1) and programmed cell death1 (PD-1) expression in the tumor, over treatment and correlate with response and survival with goal of biomarker discovery.

II. Estimate the relapse-free survival (RFS) in all enrolled subjects.

OUTLINE:

Patients receive tremelimumab IV over 1 hour and durvalumab IV over 4 hours during week 11. Between weeks 15 and 17, patients undergo liver surgery. Patients then receive durvalumab IV over 1 hour during weeks 21, 25, 29, and 33.

After completion of study treatment, patients are followed up twice a year for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed colorectal cancer with liver metastases deemed resectable by a general or liver surgeon (resectability may involve the use of ablative techniques to some but not all liver metastases); those patients with known disease outside of the liver are not eligible (except for patients with primary lesions in place that are planned for resection or nonspecific lung metastases < 1 cm)
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 10 mm with spiral computed tomography (CT) scan
* All lines of prior therapy accepted; subjects with prior hepatic or extra-hepatic resections of metastatic disease will be included
* Life expectancy of greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin < 1.5 X institutional normal limits (subjects with known Gilbert syndrome are eligible with total bilirubin < 3.0 mg/dL)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase [SGPT]) =< 3 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Known or ordered molecular testing for MSI, BRAF, and KRAS status
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients; women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause; the following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
  * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy)
* Ability to understand and the willingness to sign a written informed consent document
* Weight > 30 kg (required for flat dose-based administration of study agents)

Exclusion Criteria:

* Prior chemotherapy < 2 weeks prior to study drug treatment and treatment related adverse events that have not recovered to baseline or grade 1 (alopecia excluded); prior radiation therapy < 4 weeks prior to study drug treatment
* Patients may not be receiving any other investigational agents
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]); the following are exceptions to this criterion: a) patients with vitiligo or alopecia; b) patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement; c) any chronic skin condition that does not require systemic therapy; d) patients without active disease in the last 5 years may be included but only after consultation with the study physician; d) patients with celiac disease controlled by diet alone
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Prior exposure to T cell checkpoint inhibitor therapies, including durvalumab and tremelimumab
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, interstitial lung disease, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
* History of active primary immunodeficiency
* Women who are pregnant, which includes women with a positive pregnancy test at enrollment or prior to the administration of study medication, or breastfeeding are not allowed on study
* Receipt of a live vaccine within 30 days of study entry
* Any unresolved toxicity National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade >= 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria: a) patients with grade >= 2 neuropathy will be evaluated on a case-by-case basis after consultation with the study physician; b) patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the study physician
* Any concurrent chemotherapy, biologic, or hormonal therapy for cancer treatment, concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable
* Major surgical procedure within 28 days prior to the first dose of IP; Note: local surgery of isolated lesions for palliative intent is acceptable
* History of allogenic organ transplantation
* Known active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis [TB] testing in line with local practice), hepatitis B (known positive hepatitis B virus [HBV] surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies); patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible; patients positive for hepatitis C (hepatitis C virus [HCV]) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA)
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab + tremelimumab combination therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Overman, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 8/2016 -1/2019
Pre-assignment Details: 24 participants started and 1 participate withdrew from study( 23 participants completed the study)
Groups:
- Durvalumab/Tremelimumab: Neoadjuvant tremelimumab 75 mg IV flat dose and durvalumab 1500 mg IV flat dose given pre-operatively for 1 cycle prior to CRC liver metastases resection. Post-operative therapy was at the discretion of the treating physician, and patients were eligible to receive durvalumab 1500 mg IV every 4 weeks for 4 cycles.
Period: Overall Study
Arm/Group | Durvalumab/Tremelimumab
Started | 24
Completed | 23
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Durvalumab/Tremelimumab
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: Years] | 56 [28 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Toxicity
Description: Post-operative toxicity graded by the Clavien-Dindo classification. The Clavien Dindo Classification is used to rank the severity of a surgical complication. It is based on the type of therapy needed to correct the complication. The scale consists of several grades (Grade I, II, IIIa, IIIb, IVa, IVb and V). Grade I complications are usually mild but Grade II and higher complications are more significant.
Time Frame: 3 years
Population: 3 patients did not undergo surgical exploration because of progression of previously noted sub-centimeter lung nodules.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab/Tremelimumab
Number analyzed (Participants) | 20
Participants | 8

2. Primary Outcome: Feasibility and Safety in the Conduct of the Trial
Description: Feasibility and safety assessed by the rate of on-trial surgical resection of liver metastases, post-operative toxicity graded by the Clavien-Dindo classification, and treatment related toxicity graded by CTCAE v5. The combination was defined as feasible if at least 80% of participants could undergo resection or if between 60% and 80% could undergo resection with a positive toxicity and efficacy profile.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab/Tremelimumab
Number analyzed (Participants) | 20
Participants
  Surgical resection | 17
  Exploration, no resection | 3

3. Secondary Outcome: Treatment Related Toxicity
Description: Treatment related toxicity graded by CTCAE v5
Time Frame: 3 years
Population: Grade 3/4 treatment-related immune toxicity and postoperative grade 3/4 toxicity
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab/Tremelimumab
Number analyzed (Participants) | 23
percentage of participants | 22 [10 to 44]

4. Secondary Outcome: Pre-operative Response Rate
Description: Pre-operative response rate evaluation using RECIST v1.1. RECIST 1.1 will be used to identify measurable disease on baseline CT scans. Tumor measurements will be made upon restaging CT scans prior to surgery. No tumor measurements will take place post-operatively as the goal of therapy is no evidence of disease. Pre-surgery response will be classified into Complete Response, Partial Response, Stable Disease and Progressive Disease.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab/Tremelimumab
Number analyzed (Participants) | 23
Participants
  Stable Disease | 15
  Patial Response | 3
  Progressive disease | 5

5. Secondary Outcome: Relapse-Free Survival (RFS)
Description: The time from date of curative surgery to the time of recurrence or death
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab/Tremelimumab
Number analyzed (Participants) | 23
Months | 9.7 [1.3 to 28]

6. Secondary Outcome: Overall Survival
Description: The time from treatment to death, regardless of disease recurrence.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab/Tremelimumab
Number analyzed (Participants) | 23
months | 24.5 [16.5 to 28.4]

7. Secondary Outcome: Translational Evaluation of Various Immune-relevant Factors
Description: Tumor immune markers was evaluated using flow cytometry, Multiplex Immunofluorescence (mIF) and Immunohistochemistry (IHC) analyses, RNA sequencing, Microbial DNA isolation and 16S rRNA gene sequencing (using QIAamp DNA stool mini kit on pretreatment feacal samples)
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab/Tremelimumab
Number analyzed (Participants) | 23
Participants
  POLE mutation B | 2
  BRAF mutation | 1
  KRAS mutation | 12
  TP53 mutation | 14
  APC mutation | 11
  pMMR | 21
  dMMR | 2
  CMS1 | 0
  CMS2 | 7
  CMS3 | 4
  CMS4 | 4

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Treatment related toxicity was assessed and graded using CTCAE v5
Arm/Group | Durvalumab/Tremelimumab
All-Cause Mortality (participants affected / at risk) | 1/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 23/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Durvalumab/Tremelimumab (N=23)
Anemia (Investigations) | 2
Decreased neutrophil count (Investigations) | 2
Decreased platelet count (Investigations) | 3
Decreased white blood cells (Investigations) | 1
Hypokalemia (Investigations) | 1
Hyponatremia (Investigations) | 1
Increased alanine aminotransferase (Investigations) | 2
Increased alkaline phosphatase (Investigations) | 2
Increased aspartate aminotransferase (Investigations) | 3
Lipase increased (Investigations) | 2
Adrenal insufficiency (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 3
Serum amylase increased (Investigations) | 1
Anorexia (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Rectal hemorrhage (Gastrointestinal disorders) | 1
Chills (General disorders) | 2
Fatigue (General disorders) | 10
Fever (General disorders) | 3
Hypotention (General disorders) | 1
Anxiety (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Rash (maculo-papular) (Skin and subcutaneous tissue disorders) | 2
Rash (acneiform) (Skin and subcutaneous tissue disorders) | 2
Pruritis (Skin and subcutaneous tissue disorders) | 4
Oral mucositis (Gastrointestinal disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Insomnia (Psychiatric disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/56/NCT02754856/Prot_SAP_000.pdf